CLINICAL TRIAL: NCT01257451
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of 24 Weeks Treatment With Vildagliptin in Type 2 Diabetes Mellitus Patients ≥ 70 Years (Drug-naive or Inadequately Controlled on Oral Agents)
Brief Title: Safety and Efficacy of Galvus in Elderly Type 2 Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLAF237A23150; 2010-022658-18
Record Dates: First submitted 2010-12-06; First posted 2010-12-09 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus, Vildagliptin, Elderly Patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: Vildagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin — vildagliptin 50mg bid
  Arms: Vildagliptin
Drug: Placebo — Placebo 50mg bid
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of vildagliptin 50 mg bid in elderly patients with Type 2 Diabetes Mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* age: ≥ 70 years inclusive at Visit 1.
* patients with a confirmed diagnosis of T2DM
* HbA1c of ≥ 7% and ≤10.0% by central laboratory at Visit 1 and assessed by the investigator to be inadequately controlled
* body mass index (BMI) in the range of 19-45kg/m2

Exclusion Criteria:

* FPG ≥ 270 mg/dL (≥ 15.0 mmol/L)
* previous or current participation in any vildagliptin clinical study.
* history of hypersensitivity to DPP-4 inhibitors.
* concurrent medical condition that may interfere with the interpretation of efficacy and safety data during the study.
* donation of blood or significant blood loss equaling to at least one unit of blood within the past 2 weeks of start of study or a blood transfusion within the past 12 weeks or planned regular transfusions during the study period Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 431 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the proportion of vildagliptin treated patients achieving HbA1c reduction and/or proportion reaching investigator defined target HbA1c relative to placebo | 24 weeks

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of vildagliptin in elderly patients with T2DM who are drug-naive or inadequately controlled with oral antidiabetic drugs (OADs) including physical exam, vital sign, hematology, chemistry and electrocardiogram. | 24 weeks
To evaluate the proportion of vildagliptin treated patients achieving fasting plasma glucose (FPG) reduction relative to placebo | 24 weeks
To assess the responder rates of patients treated with vildagliptin as compared to placebo | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals Corporation, Study Director — Novartis Pharmaceuticals
Locations (46):
- Belgium (7):
  - Novartis Investigative Site, Wichelen, Belgium
  - Novartis Investigative Site, Buizingen
  - Novartis Investigative Site, De Pinte
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Mouscron
  - Novartis Investigative Site, Nazareth
  - Novartis Investigative Site, Oostham
- Bulgaria (7):
  - Novartis Investigative Site, Blagoevgrad, Bulgaria
  - Novartis Investigative Site, Dimitrovgrad, Bulgaria
  - Novartis Investigative Site, Plovdiv, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Varna, Bulgaria
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- Finland (3):
  - Novartis Investigative Site, Lahti, Suomi
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Oulu
- Germany (13):
  - Novartis Investigative Site, Münster, Germany
  - Novartis Investigative Site, Völlkingen, Germany
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Beckum
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Eisleben Lutherstadt
  - Novartis Investigative Site, Falkensee
  - Novartis Investigative Site, Lichtenfels
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mammendorf
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Sulzbach-Rosenberg
  - Novartis Investigative Site, Wetter
- Slovakia (7):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Ľubochňa, Slovak Republic
  - Novartis Investigative Site, Levice, Slovakia
  - Novartis Investigative Site, Nové Zámky, Slovakia
  - Novartis Investigative Site, Pie¿¿any, Slovakia
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Ružomberok
- Spain (4):
  - Novartis Investigative Site, Alicante, Alicante
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Centelles, Barcelona
  - Novartis Investigative Site, Alzira, Valencia
- United Kingdom (5):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Stevenage
  - Novartis Investigative Site, Wiltshire

REFERENCES:
- [Derived] Strain WD, Lukashevich V, Kothny W, Hoellinger MJ, Paldanius PM. Individualised treatment targets for elderly patients with type 2 diabetes using vildagliptin add-on or lone therapy (INTERVAL): a 24 week, randomised, double-blind, placebo-controlled study. Lancet. 2013 Aug 3;382(9890):409-416. doi: 10.1016/S0140-6736(13)60995-2. Epub 2013 May 23. PMID 23706759